CLINICAL TRIAL: NCT02565381
Title: The QUIT Smoking Study: A Pilot Randomized Controlled Trial of Financial Incentives, Text Messaging, and Usual Care to Help Homeless Smokers Quit Smoking
Brief Title: A Pilot Randomized Controlled Trial of Financial Incentives, Text Messaging, and Usual Care for Homeless Smokers
Acronym: QUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Travis Paul Baggett, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001300; K23DA034008 (NIH)
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (N=25) (Active Comparator): * Transdermal nicotine patch
  * In-person smoking cessation counseling
  Interventions: Drug: Transdermal nicotine patch; Behavioral: In-person smoking cessation counseling
- Financial rewards (N=25) (Experimental): * Transdermal nicotine patch
  * In-person smoking cessation counseling
  * Contingent financial rewards for smoking abstinence
  Interventions: Drug: Transdermal nicotine patch; Behavioral: In-person smoking cessation counseling; Behavioral: Contingent financial rewards for smoking abstinence
- Text messaging (N=25) (Experimental): * Transdermal nicotine patch
  * In-person smoking cessation counseling
  * Text messages to support smoking abstinence
  Interventions: Drug: Transdermal nicotine patch; Behavioral: In-person smoking cessation counseling; Behavioral: Text messages to support smoking abstinence

INTERVENTIONS:
Drug: Transdermal nicotine patch — * ≥10 cigarettes per day: nicotine 21mg/24hr patch daily x 6 weeks, then nicotine 14mg/24hr patch daily x 2 weeks
  * <10 cigarettes per day: nicotine 14mg/24hr patch daily x 8 weeks
  Other Names: Nicotine
Behavioral: In-person smoking cessation counseling — - One-on-one 15-minute counseling sessions once per week for 8 weeks
Behavioral: Contingent financial rewards for smoking abstinence — - Escalating-value financial rewards for smoking abstinence, verified by exhaled carbon monoxide <8ppm
  Other Names: Contingency management
  Arms: Financial rewards (N=25)
Behavioral: Text messages to support smoking abstinence — - 1-5 text messages per day starting up to 2 weeks before the quit date and continuing until 6 weeks after the quit date, delivered by SmokefreeTXT
  Arms: Text messaging (N=25)

SUMMARY:
The QUIT (Quitting with Usual Care, Incentives, and Technology) Smoking Study is a 3-arm pilot randomized controlled trial that will test the effect of 2 different experimental smoking cessation interventions relative to a control condition in homeless cigarette smokers. All participants will receive free transdermal nicotine patches and weekly in-person smoking cessation counseling. In addition, participants randomized to the first experimental condition will receive financial rewards for biochemically-verified smoking abstinence, and participants randomized to the second experimental condition will be enrolled in a text messaging program to support smoking abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Proficient in English, assessed with items asking about native language and self-reported comfort communicating in English among non-native speakers.
* Age ≥18 years old, assessed by self-report and verified by date of birth.
* Has smoked ≥100 cigarettes and currently smokes ≥5 cigarettes per day, verified by an exhaled carbon monoxide level of ≥8 ppm.
* Ready to try quitting smoking within the next month.
* Currently homeless, assessed by self-report and defined as usually staying in an emergency shelter, transitional shelter, abandoned building, place of business, car or other vehicle, church or mission, hotel or motel, or anywhere outside during the past 7 days. Additionally, individuals will be considered currently homeless if they usually stayed in somebody else's house, apartment/condominium, or room in the past 7 days because of not having their own place to stay.

Exclusion Criteria:

* Currently pregnant, assessed by a urine pregnancy test conducted on all premenopausal biologic females who have not had a hysterectomy, or planning to become pregnant in the next 2 months.
* Past 30-day use of nicotine replacement therapy, bupropion, or varenicline for smoking cessation, assessed by self-report. Use of bupropion for reasons other than to quit smoking (e.g. depression) is permissible.
* Prior serious adverse reaction to the nicotine patch, defined as any reaction that was life-threatening or required hospitalization.
* Heart attack or chest pain within the past 2 weeks.
* Inability to read a sentence written at a Flesch-Kincaid grade level of 4.
* Inability to provide informed consent, assessed with knowledge questions about the material presented during the informed consent process that individuals must correctly answer before providing informed consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis P Baggett, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Boston Health Care for the Homeless Program, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Baggett TP, McGlave C, Kruse GR, Yaqubi A, Chang Y, Rigotti NA. SmokefreeTXT for Homeless Smokers: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 4;7(6):e13162. doi: 10.2196/13162. PMID 31165717
- [Derived] Baggett TP, Yaqubi A, Berkowitz SA, Kalkhoran SM, McGlave C, Chang Y, Campbell EG, Rigotti NA. Subsistence difficulties are associated with more barriers to quitting and worse abstinence outcomes among homeless smokers: evidence from two studies in Boston, Massachusetts. BMC Public Health. 2018 Apr 10;18(1):463. doi: 10.1186/s12889-018-5375-z. PMID 29631559
- [Derived] Baggett TP, Chang Y, Yaqubi A, McGlave C, Higgins ST, Rigotti NA. Financial Incentives for Smoking Abstinence in Homeless Smokers: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2018 Nov 15;20(12):1442-1450. doi: 10.1093/ntr/ntx178. PMID 29059442

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants (N=8) enrolled in the study but did not return for randomization.
Groups:
- Control (N=25): * Transdermal nicotine patch
  * In-person smoking cessation counseling
  Transdermal nicotine patch: - ≥10 cigarettes per day: nicotine 21mg/24hr patch daily x 6 weeks, then nicotine 14mg/24hr patch daily x 2 weeks
  - <10 cigarettes per day: nicotine 14mg/24hr patch daily x 8 weeks
  In-person smoking cessation counseling: - One-on-one 15-minute counseling sessions once per week for 8 weeks
- Financial Rewards (N=25): * Transdermal nicotine patch
  * In-person smoking cessation counseling
  * Contingent financial rewards for smoking abstinence
  Transdermal nicotine patch: - ≥10 cigarettes per day: nicotine 21mg/24hr patch daily x 6 weeks, then nicotine 14mg/24hr patch daily x 2 weeks
  - <10 cigarettes per day: nicotine 14mg/24hr patch daily x 8 weeks
  In-person smoking cessation counseling: - One-on-one 15-minute counseling sessions once per week for 8 weeks
  Contingent financial rewards for smoking abstinence: - Escalating-value financial rewards for smoking abstinence, verified by exhaled carbon monoxide <8ppm
- Text Messaging (N=25): * Transdermal nicotine patch
  * In-person smoking cessation counseling
  * Text messages to support smoking abstinence
  Transdermal nicotine patch: - ≥10 cigarettes per day: nicotine 21mg/24hr patch daily x 6 weeks, then nicotine 14mg/24hr patch daily x 2 weeks
  - <10 cigarettes per day: nicotine 14mg/24hr patch daily x 8 weeks
  In-person smoking cessation counseling: - One-on-one 15-minute counseling sessions once per week for 8 weeks
  Text messages to support smoking abstinence: - 1-5 text messages per day starting up to 2 weeks before the quit date and continuing until 6 weeks after the quit date, delivered by SmokefreeTXT
Period: Overall Study
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Started | 25 | 25 | 25
Completed | 24 | 25 | 24
Not Completed | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25) | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (9.6) | 48.1 (8.5) | 46.1 (9.2) | 46.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 15 | 41
  Male | 11 | 13 | 10 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 2 | 13
  Not Hispanic or Latino | 20 | 19 | 23 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 3 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 11 | 11 | 31
  White | 10 | 11 | 10 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 1 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 25 | 75
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Score range is 0-10, with higher scores indicating greater nicotine dependence.
  units on a scale | 5.1 (1.8) | 5.1 (1.9) | 4.9 (2.0) | 5.0 (1.9)
Quitting confidence [Mean (Standard Deviation); unit: units on a scale] — 1-10 visual scale of confidence to quit, with higher scores indicating greater confidence to quit smoking.
  units on a scale | 6.8 (2.2) | 6.4 (2.5) | 5.9 (2.4) | 6.4 (2.4)
Quitting importance [Mean (Standard Deviation); unit: units on a scale] — 1-10 visual scale of importance of quitting, with higher scores indicating greater importance of quitting smoking.
  units on a scale | 8.8 (1.5) | 8.5 (2.1) | 8.9 (1.6) | 8.8 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biochemically-verified Smoking Abstinence, Assessed 14 Times Over 8 Weeks
Description: The primary outcome is a repeated-measures assessment of smoking abstinence, defined as an exhaled carbon monoxide <8ppm and assessed 14 times over the 8-week study period (3 times/week for the first 2 weeks, 2 times/week for the next 2 weeks, and once every week for the last 4 weeks)
Time Frame: Point-in-time abstinence assessed in a repeated fashion 14 times over the 8-week study period
Population: Participants with missing data at a given time point were assumed non-abstinent at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 25 | 25 | 25
Participants
  Day 3 | 3 | 10 | 3
  Day 5 | 0 | 9 | 1
  Day 7 | 4 | 15 | 3
  Day 10 | 4 | 15 | 2
  Day 12 | 5 | 17 | 4
  Day 14 | 4 | 15 | 4
  Day 17 | 3 | 13 | 4
  Day 21 | 2 | 14 | 3
  Day 24 | 2 | 17 | 5
  Day 28 | 4 | 12 | 2
  Day 35 | 4 | 8 | 3
  Day 42 | 4 | 11 | 2
  Day 49 | 3 | 11 | 1
  Day 56 | 2 | 12 | 4

2. Secondary Outcome: Percentage of Visits Abstinent of Smoking
Description: Percentage of 14 assessment visits at which a participant is abstinent of smoking, defined as an exhaled carbon monoxide level <8ppm.
Time Frame: 8 weeks
Population: Participants with missing data at a given time point were assumed non-abstinent at that time point.
Measure: Mean (Standard Deviation); unit: percentage of visits
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 25 | 25 | 25
percentage of visits | 12.6 (22.1) | 51.1 (32.8) | 11.7 (21.9)

3. Secondary Outcome: Smoking Abstinence at End of Study
Description: Point-prevalence smoking abstinence, defined as an exhaled carbon monoxide level <8ppm, at the 14th (final) study visit.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 25 | 25 | 25
Participants | 2 | 12 | 4

4. Secondary Outcome: Change in Cigarette Consumption
Description: Changes in the average number of cigarettes per day relative to baseline, defined by self-report and repeatedly assessed at the 8 assessment visits occurring on Fridays.
Time Frame: Once per week for 8 weeks
Population: Participants with missing data at a given time point are excluded from calculation of mean changes in cigarette consumption for that time point.
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 24 | 25 | 24
Cigarettes per day
  Week 1: number analyzed (Participants) | 19 | 22 | 18
  Week 1 | -5.3 (6.1) | -8.5 (6.0) | -6.0 (7.2)
  Week 2: number analyzed (Participants) | 17 | 18 | 17
  Week 2 | -6.7 (5.8) | -8.6 (6.8) | -7.5 (6.8)
  Week 3: number analyzed (Participants) | 14 | 15 | 16
  Week 3 | -8.5 (5.4) | -12.3 (10.2) | -7.7 (7.2)
  Week 4: number analyzed (Participants) | 16 | 17 | 16
  Week 4 | -8.0 (5.6) | -11.1 (6.9) | -9.5 (7.2)
  Week 5: number analyzed (Participants) | 13 | 13 | 15
  Week 5 | -9.4 (6.4) | -10.2 (7.2) | -7.9 (7.0)
  Week 6: number analyzed (Participants) | 14 | 14 | 13
  Week 6 | -6.2 (4.2) | -10.4 (6.7) | -5.4 (5.2)
  Week 7: number analyzed (Participants) | 15 | 14 | 16
  Week 7 | -8.6 (6.4) | -10.1 (7.2) | -8.1 (8.0)
  Week 8: number analyzed (Participants) | 16 | 17 | 16
  Week 8 | -8.7 (5.9) | -7.9 (5.5) | -5.4 (3.7)

5. Secondary Outcome: Change in Behavioral Health
Description: Past-month drug use severity (score range 0-1), past-month alcohol use severity (score range 0-1), and past-month psychiatric severity (0-1) were each assessed with the Addiction Severity Index (ASI) - 5th Edition, at baseline and at the 10th and 14th study visits. For each ASI measure, higher scores represent greater drug, alcohol, or psychiatric severity. Changes in ASI scores between baseline and 4 or 8 weeks can range from -1 to +1. When interpreting changes in scores, negative values indicate decreases in scores from baseline to 4 or 8 weeks, and positive values indicate increases in scores from baseline to 4 or 8 weeks.
Time Frame: 4 weeks and 8 weeks
Population: Participants with missing data at a particular time point are excluded from calculation of mean change in ASI scores at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 24 | 25 | 24
units on a scale
  ASI alcohol 4 wk change | -0.02 (0.12) | -0.04 (0.10) | -0.09 (0.13)
  ASI alcohol 8 wk change | -0.01 (0.13) | 0.01 (0.13) | -0.04 (0.14)
  ASI drug 4 wk change | -0.02 (0.08) | -0.04 (0.07) | -0.03 (0.09)
  ASI drug 8 wk change | -0.02 (0.08) | -0.01 (0.08) | 0 (0.09)
  ASI psychiatric 4 wk change | -0.06 (0.22) | -0.04 (0.13) | -0.01 (0.20)
  ASI psychiatric 8 wk change | -0.04 (0.21) | 0.08 (0.17) | -0.04 (0.16)

6. Secondary Outcome: Study Visit Attendance
Description: Percentage of 14 assessment visits attended.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of visits
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 25 | 25 | 25
percentage of visits | 65.4 (32.2) | 71.1 (24.3) | 65.7 (27.0)

7. Secondary Outcome: Counseling Visit Attendance
Description: Percentage of 8 counseling visits attended.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of visits
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 25 | 25 | 25
percentage of visits | 17.0 (21.3) | 10.5 (12.8) | 17.0 (21.0)

8. Secondary Outcome: Nicotine Patch Use
Description: Days of nicotine replacement therapy use in past week, repeatedly measured at the 8 assessment visits occurring on Fridays.
Time Frame: 8 weeks
Population: Participants with missing data at a given time point were excluded from calculation of mean past-week patch use at that time point.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 24 | 25 | 24
Days
  Week 1: number analyzed (Participants) | 19 | 21 | 17
  Week 1 | 3.7 (2.7) | 4.1 (2.6) | 4.5 (2.9)
  Week 2: number analyzed (Participants) | 16 | 18 | 17
  Week 2 | 4.9 (2.8) | 4.5 (2.6) | 4.5 (2.9)
  Week 3: number analyzed (Participants) | 14 | 15 | 16
  Week 3 | 4.4 (2.9) | 4.9 (2.2) | 4.9 (2.9)
  Week 4: number analyzed (Participants) | 16 | 18 | 17
  Week 4 | 4.3 (3.0) | 3.6 (2.8) | 4.4 (2.8)
  Week 5: number analyzed (Participants) | 13 | 13 | 14
  Week 5 | 4.4 (2.7) | 4.6 (2.8) | 4.9 (2.5)
  Week 6: number analyzed (Participants) | 15 | 14 | 13
  Week 6 | 3.5 (2.8) | 4.0 (3.0) | 4.1 (2.7)
  Week 7: number analyzed (Participants) | 15 | 14 | 16
  Week 7 | 4.3 (2.8) | 4.6 (2.5) | 3.8 (2.6)
  Week 8: number analyzed (Participants) | 17 | 19 | 17
  Week 8 | 3.6 (3.1) | 3.9 (2.9) | 2.7 (2.9)

9. Other Pre Specified Outcome: Recruitment Time
Description: Total time to recruit, enroll, and randomize 75 study participants.
Time Frame: Until target number of participants is reached; anticipate ~6 months
Measure: Number; unit: months
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 25 | 25 | 25
months | 6 | 6 | 6

10. Other Pre Specified Outcome: Mobile Phone Retention
Description: Percentage of participants who still have their mobile phone at the end of the study.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 25 | 25 | 25
Participants | 13 | 15 | 10

11. Other Pre Specified Outcome: Use of Text Messaging Program
Description: Text messaging group only: number who enrolled in SmokefreeTXT, number who replied to query texts sent by SmokefreeTXT.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
Number analyzed (Participants) | 0 | 0 | 25
Participants
  Enrolled in SmokefreeTXT |  |  | 22
  Replied to texts from SmokefreeTXT |  |  | 7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 8-week study period for each participant.
Description: Participants were asked about adverse events at each of the 14 follow-up visits over 8 weeks.
Arm/Group | Control (N=25) | Financial Rewards (N=25) | Text Messaging (N=25)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 0/25 | 5/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=25) (N=25) | Financial Rewards (N=25) (N=25) | Text Messaging (N=25) (N=25)
Nausea/vomiting (Gastrointestinal disorders) | 0 | 0 | 2 — Nausea or vomiting correlated with nicotine patch use
Rash at nicotine patch site (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Rash at nicotine patch site
Dizziness (Nervous system disorders) | 0 | 0 | 2 — Dizziness correlated with nicotine patch use
Sweating (General disorders) | 0 | 0 | 2 — Sweatiness correlated with nicotine patch use
Headache (General disorders) | 0 | 0 | 1 — Headache correlated with nicotine patch use
Fatigue (General disorders) | 0 | 0 | 1 — Fatigue correlated with nicotine patch use

LIMITATIONS AND CAVEATS:
Small sample size; short duration of follow-up; primary outcome based exclusively on exhaled carbon monoxide measurement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes